CLINICAL TRIAL: NCT06363851
Title: A Phase 1 Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Ascending Doses of Kylo-11 in Healthy Subjects
Brief Title: Single-ascending Dose Study of Kylo-11 in Healthy Subjects
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Kylonova (Xiamen) Biopharma co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Kylo-11-I-C01
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-05

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kylo-11 (Experimental): Single ascending doses of Kylo-11 administered subcutaneously (SC).
  Interventions: Drug: Kylo-11
- Placebo (Placebo Comparator): Administered SC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Kylo-11 — Administered SC.
  Arms: Kylo-11
Drug: Placebo — Administered SC.
  Arms: Placebo

SUMMARY:
This is a first-in-human, randomized, double-blind, placebo-controlled, single ascending dose study in healthy volunteers. Kylo-11 will be evaluated in approximately 60 subjects to assess safety, tolerability, pharmacokinetics and pharmacodynamic effects.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 to 55 years old, inclusive;
* Body mass index (BMI) between 19 kg/m2 and 30 kg/m2, inclusive;
* Protocol-defined elevated serum Lp(a) level;
* Female subjects must not be able to get pregnant and male subjects must agree to adhere to contraception restrictions;
* Willing to comply with protocol required visits and assessments, and provide written informed consent.

Exclusion Criteria:

* History or evidence of a clinically significant disorder, condition or disease;
* Received an investigational drug, vaccine or device within 3 months before dosing;
* History of evidence of malignant tumor or Gilbert syndrome;
* Positive screen of Hepatitis B surface antigen, hepatitis C virus, human immunodeficiency virus or syphilis infection;
* History of alcohol abuse within 12 months before dosing;
* History of drug abuse within 3 months before screening;
* History of blood donations or blood loss of 400 ml and more within 3 months before dosing;
* History of stroke or myocardial infarction within 6 months before sceening;
* Pregnant or breast-feeding women;
* Other exclusion criteria applied per protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-16 (Actual); Primary Completion 2025-06-17 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | up to Week 24

SECONDARY OUTCOMES:
Incidence of adverse events | up to week 48
Pharmacokinetics (PK) parameter of maximum observed concentration (Cmax) | up to Week 48
PK parameter of time of maximum observed concentration (Tmax) | up to Week 48
PK parameter of area under the concentration time curve (AUC) | up to Week 48
Change in serum Lp(a) over time | up to Week 48
Percent change in serum Lp(a) over time | up to Week 48

CONTACTS AND LOCATIONS:
Locations (1):
- Chengdu Xinhua Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No